CLINICAL TRIAL: NCT05149313
Title: A Randomised, Double-Blind, Placebo-Controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of Lebrikizumab in Combination With Topical Corticosteroids in Adult and Adolescent Patients With Moderate-To-Severe Atopic Dermatitis That Are Not Adequately Controlled With Cyclosporine or For Whom Cyclosporine is Not Medically Advisable.
Brief Title: A Study of Lebrikizumab in Combination With Topical Corticosteroids in Patients With Atopic Dermatitis (AD) That Are Not Adequately Controlled With or Are Non-eligible for Cyclosporine
Acronym: ADvantage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-17923-30; 2021-002967-23 (EudraCT Number)
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Dermatitis, Atopic; Eczema
Keywords: Topical Corticosteroids; Cyclosporine
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lebrikizumab (Experimental): Lebrikizumab administered subcutaneously (SC), participants will receive 2 injections of lebrikizumab 250 mg at Baseline and Week 2, followed by 1 injection of lebrikizumab 250 milligram (mg) once every two weeks (Q2W) in the induction period up to week 16. Participants who received lebrikizumab 250 mg Q2W during the Induction Period will continue to receive lebrikizumab 250 mg Q2W during the Maintenance Period. In order to maintain the double blind, participants from the lebrikizumab 250 mg Q2W arm will be administered a second injection of blinded placebo during Week 16 and Week 18. From Week 20 up to Week 52, all participants will receive 1 injection of lebrikizumab 250 mg Q2W in Open-label maintenance period.
  Interventions: Biological: Lebrikizumab
- Lebrikizumab-matching Placebo (Placebo Comparator): Lebrikizumab-matching Placebo administered SC, 250 mg dose, Q2W in the induction period for 16 weeks. Participants will receive 2 injections of lebrikizumab 250 mg at Week 16 and Week 18 followed by 1 injection of lebrikizumab 250 mg Q2W from Week 20 up to Week 52 in Open-label maintenance period.
  Interventions: Drug: Lebrikizumab-matching Placebo

INTERVENTIONS:
Biological: Lebrikizumab — Lebrikizumab solution for injection administered subcutaneously.
  Arms: Lebrikizumab
Drug: Lebrikizumab-matching Placebo — Matching Placebo solution for injection administered subcutaneously.
  Arms: Lebrikizumab-matching Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of lebrikizumab compared with placebo in participants not adequately controlled with cyclosporine or for whom cyclosporine is not medically advisable up to Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Adults and adolescents (aged greater than or equal to (>=) 12 to <18 years at the time of Informed Consent Form (ICF)/Informed Assent Form (IAF) and weighing >=40 kilograms).
* Chronic AD that has been present for >=1 year before the Screening visit.
* EASI score >=16 at the Baseline Visit.
* IGA score >=3 (moderate) (scale of 0 [clear] to 4 [severe]) at the Baseline visit.
* >=10% BSA of AD involvement at the Baseline visit.
* Inadequate response to existing topical medications
* Failure to cyclosporine or non-medically advisable to receive/continue receiving cyclosporine
* Signed ICF (and informed assent for adolescents as required)

Exclusion Criteria:

* Treatment with TCS within 1 week before the Baseline visit.
* Treatment with topical calcineurin inhibitors, phosphodiesterase-4 inhibitors such as crisaborole, or cannabinoids within 2 week before the Baseline visit.
* Treatment with interleukin 4 (IL-4) or interleukin 13 (IL-13) antagonists biological therapies before the Baseline visit. Exception: previous treatment with dupilumab will be allowed in a subset of patients
* Treatment with immunosuppressive/immunomodulating drugs, phototherapy and photochemotherapy within 4 weeks before the Baseline visit
* Uncontrolled chronic disease that might require bursts of oral corticosteroids
* Serious, opportunistic, chronic or recurring infections within 3 months of Screening or before randomization
* Current or chronic infection with hepatitis B virus, current infection with hepatitis C virus, known liver cirrhosis and/or chronic hepatitis of any etiology
* Known or suspected history of immunosuppression, history of HIV infection or positive HIV serology at Screening
* Any clinically significant laboratory test results obtained at the Screening visit
* Presence of skin comorbidities that may interfere with study assessments
* Have had an important side effect to TCS that would prevent further use.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (48):
- Alm Site 1, Graz, Austria
- Alm Site 2, Ghent, Belgium
- France (9):
  - Alm Site 14, Bordeaux
  - Alm Site 17, Le Mans
  - Alm Site 19, Lille
  - Alm Site 20, Lille
  - Alm Site 13, Martigues
  - Alm Site 16, Nantes
  - Alm Site 15, Nice
  - Alm Site 18, Pierre-Bénite
  - Alm Site 12, Reims
- Germany (9):
  - Alm Site 28, Bad Bentheim
  - Alm Site 30, Berlin
  - Alm Site 24, Blankenfelde
  - Alm Site 32, Bonn
  - Alm Site 31, Frankfurt
  - Alm Site 27, Göttingen
  - Alm Site 26, Hamburg
  - Alm Site 29, Kiel
  - Alm Site 25, Marburg
- Netherlands (3):
  - Alm Site 34, Bergen op Zoom
  - Alm Site 33, Rotterdam
  - Alm Site 35, Utrecht
- Poland (13):
  - Alm Site 45, Bialystok
  - Alm Site 43, Chorzów
  - Alm Site 38, Katowice
  - Alm Site 41, Krakow
  - Alm Site 46, Krakow
  - Alm Site 37, Lodz
  - Alm Site 39, Lublin
  - Alm Site 48, Ostrowiec Świętokrzyski
  - Alm Site 44, Rzeszów
  - Alm Site 36, Szczecin
  - Alm Site 42, Warsaw
  - Alm Site 47, Warsaw
  - Alm Site 40, Wroclaw
- Spain (9):
  - Alm Site 10, Alicante
  - Alm Site 3, Badalona
  - Alm Site 6, Barcelona
  - Alm Site 8, Barcelona
  - Alm Site 4, Bilbao
  - Alm Site 5, Madrid
  - Alm Site 11, Mieres
  - Alm Site 7, Seville
  - Alm Site 9, Zaragoza
- United Kingdom (3):
  - Alm Site 23, Poole
  - Alm Site 22, Salford
  - Alm Site 21, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 54 sites in Austria, Belgium, France, Germany, Italy, Netherlands, Poland, Spain, and United Kingdom. Randomization was stratified by previous use of dupilumab, age (adolescent participants aged >=12 to < 18 years comprises 11.8% of the overall population compared to adults aged >=18 years) and baseline disease severity (IGA 3 vs 4).
Pre-assignment Details: A total of 368 participants were screened, of which 331 participants were randomized into 2 treatment arms (Lebrikizumab and Placebo). The study has 2 treatment periods: a 16-week double-blind Induction Period and 36-week open-label Maintenance Period.
Groups:
- Double-blind Induction Period: Lebrikizumab +TCS: Participants received loading dose of lebrikizumab 500 milligrams (mg) subcutaneous (SC) injection at Day 1 (Baseline) and Week 2 followed by lebrikizumab 250 mg SC injection once every two weeks (Q2W) for up to 16 weeks concomitantly with topical corticosteroids (TCS) in the double-blind induction period.
- Double-blind Induction Period: Placebo +TCS: Participants received lebrikizumab-matched placebo SC injection, Q2W for up to 16 weeks concomitantly with TCS in the double-blind induction period.
- Open-label Maintenance Period: Lebrikizumab to Lebrikizumab: Participants who received lebrikizumab 250 mg Q2W during the Double-blind Induction Period continued to receive lebrikizumab 250 mg, Q2W during the 36-week Maintenance Period.
- Open-label Maintenance Period: Placebo to Lebrikizumab: During Maintenance Period, participants who received placebo Q2W during the Induction Period received loading doses of lebrikizumab (500 mg) at Weeks 16 and 18. From Week 20 onward, the participants received 1 injection of lebrikizumab 250mg Q2W.
Period: Double-blind Induction Period (16-weeks)
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS | Open-label Maintenance Period: Lebrikizumab to Lebrikizumab | Open-label Maintenance Period: Placebo to Lebrikizumab
Started | 220 | 111 | 0 | 0
Completed | 212 | 100 | 0 | 0
Not Completed | 8 | 11 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Period: Open-label Maintenance Period (36 Weeks)
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS | Open-label Maintenance Period: Lebrikizumab to Lebrikizumab | Open-label Maintenance Period: Placebo to Lebrikizumab
Started | 0 | 0 | 212 | 100
Completed | 0 | 0 | 180 | 87
Not Completed | 0 | 0 | 32 | 13
Not completed — Adverse Event | 0 | 0 | 7 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 14 | 7
Not completed — Lack of Efficacy | 0 | 0 | 6 | 5
Not completed — Lost to Follow-up | 0 | 0 | 4 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants and were analyzed under the treatment group as randomized.
Groups:
- Double-blind Induction Period: Lebrikizumab +TCS: Participants received loading dose of lebrikizumab 500 mg SC injection at Day 1 (Baseline) and Week 2 followed by lebrikizumab 250 mg SC injection Q2W for up to 16 weeks concomitantly with TCS in the double-blind induction period.
- Total: Total of all reporting groups
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS | Total
Number analyzed (Participants) | 220 | 111 | 331
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (14.85) | 34.1 (15.24) | 33.8 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 56 | 156
  Male | 120 | 55 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 28
  Not Hispanic or Latino | 197 | 93 | 290
  Unknown or Not Reported | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 206 | 104 | 310
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved Eczema Area and Severity Index (EASI) 75 (>=75% Reduction From Baseline in EASI Score) at Week 16
Description: The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The area of AD involvement on each of the 4 anatomic regions was assessed as a percentage by body area: 0=no eruption, 1=1% to 9%, 2=10% to 29%, 3=30% to 49%, 4=50% to 60%, 5=70% to 80% and 6=90% to 100%. The composite index with total score ranged from 0 to 72, where higher scores indicates more severe and or extensive disease.
Time Frame: At Week 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Number; unit: Percentage of participants
Groups:
- Double-blind Induction Period: Lebrikizumab +TCS: Participants received loading dose of lebrikizumab 500 mg SC injection at Day 1 (Baseline) and Week 2 followed by lebrikizumab 250 mg SC injection once Q2W for up to 16 weeks concomitantly with TCS in the double-blind induction period.
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Percentage of participants | 68.4 | 40.8
Statistical Analysis 1: Comparison: Double-blind Induction Period: Lebrikizumab +TCS vs Double-blind Induction Period: Placebo +TCS; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentages = 27.88, 95% CI 2-sided [15.63 to 40.14]

2. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved Investigator Global Assessment (IGA) Score of 0 or 1 and 2-point Improvement at Week 16
Description: The IGA is an instrument used to globally rate the severity of the participants AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting (minimal, palpable induration and significant induration). Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear).
Time Frame: At Week 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Percentage of participants | 42.0 | 24.5
Statistical Analysis 1: Comparison: Double-blind Induction Period: Lebrikizumab +TCS vs Double-blind Induction Period: Placebo +TCS; Test type: Superiority; p = 0.0052, Cochran-Mantel-Haenszel; Difference in percentages = 17.80, 95% CI 2-sided [7.03 to 28.57]

3. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved a 4-point Improvement in Pruritus Numeric Rating Score (NRS) at Week 16
Description: The Pruritus NRS is an 11-point scale used by participants to rate their worst pruritus (itch) severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable. Higher score indicates more severity.
Time Frame: At Week 16
Population: FAS included all randomized participants with the Baseline score >=4. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 199 | 102
Percentage of participants | 49.9 | 29.7
Statistical Analysis 1: Comparison: Double-blind Induction Period: Lebrikizumab +TCS vs Double-blind Induction Period: Placebo +TCS; Test type: Superiority; p = 0.0114, Cochran-Mantel-Haenszel; Difference in percentages = 18.15, 95% CI 2-sided [5.47 to 30.83]

4. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved EASI 75 (>=75% Reduction From Baseline in EASI Score) at Weeks 2, 4, 8, and 12
Description: The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The area of AD involvement on each of the 4 anatomic regions was assessed as a percentage by body area: 0=no eruption, 1=1% to 9%, 2=10% to 29%, 3=30% to 49%, 4=50% to 60%, 5=70% to 80% and 6=90% to 100%. The composite index with total score ranged from 0 to 72, where higher scores indicates more severe and or extensive disease. Percentage of participants who achieved EASI 75 (>=75% reduction from baseline in EASI score) at Weeks 2, 4, 8, and 12 were reported
Time Frame: At Weeks 2, 4, 8, and12
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Percentage of participants
  At Week 2 | 9.7 | 6.3
  At Week 4 | 28.3 | 19.2
  At Week 8 | 54.9 | 31.5
  At Week 12 | 64.9 | 41.1

5. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved EASI 90 (>=90% Reduction From Baseline in EASI Score) at Weeks 2, 4, 8, 12 and 16
Description: The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The area of AD involvement on each of the 4 anatomic regions was assessed as a percentage by body area: 0=no eruption, 1=1% to 9%, 2=10% to 29%, 3=30% to 49%, 4=50% to 60%, 5=70% to 80% and 6=90% to 100%. The composite index with total score ranged from 0 to 72, where higher scores indicates more severe and or extensive disease.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Percentage of participants
  At Week 2 | 1.5 | 0.9
  At Week 4 | 15.8 | 6.4
  At Week 8 | 28.9 | 10.6
  At Week 12 | 42.1 | 21.0
  At Week 16 | 42.9 | 20.8

6. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved EASI 50 (>=50% Reduction From Baseline in EASI Score) at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 5
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Percentage of participants
  At Week 2 | 30.8 | 23.4
  At Week 4 | 58.9 | 46.0
  At Week 8 | 75.2 | 59.3
  At Week 12 | 80.3 | 68.0
  At Week 16 | 82.6 | 65.3

7. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved a 4-point Improvement in Dermatology Life Quality Index (DLQI) at Weeks 2, 4, 8, 12 and 16
Description: The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's quality of life (QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question was scored on a 4-point scale (ranged from 0 to 3) where, 0 = not at all, 1= a little, 2= a lot, 3= very much, giving a total score ranging from 0 (not at all) to 30 (very much). A high score is indicative of a poor QoL.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: FAS included all randomized participants with Baseline DLQI score of >=4. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 180 | 90
Percentage of participants
  At Week 2 | 52.8 | 57.1
  At Week 4 | 66.1 | 61.9
  At Week 8 | 70.5 | 56.1
  At Week 12 | 73.1 | 59.6
  At Week 16 | 78.0 | 69.6

8. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved a 4-point Improvement in Children's Dermatology Life Quality Index (CDLQI) at Weeks 2, 4, 8, 12 and 16
Description: The CDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI to measure the impact of AD disease on QoL in children during the previous week. Each question is scored as follows: 0=not at all or unanswered, 1 = only a little, 2 = quite a lot and 3 = very much. Question 7 has an added possible response, which was scored as 3. CDLQI equals the sum of the score of each question, ranged from 0 (no impact of skin disease on QoL) to 30 (maximum impact on QoL). Higher scores indicate higher impact on QoL.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: FAS included all randomized participants with Baseline Score >= 4. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 22 | 8
Percentage of participants
  At Week 2 | 90.9 | 100
  At Week 4 | 68.2 | 62.5
  At Week 8 | 90.9 | 100
  At Week 12 | 95.5 | 100
  At Week 16 | 93.1 | 100

9. Secondary Outcome: Double-blind Induction Period: Percentage of Participants Who Achieved a 4- Point Improvement in Skin Pain NRS at Week 16
Description: The Skin Pain NRS is an 11-point scale completed by participants to rate their worst skin pain (example, discomfort or soreness) severity over the past 24 hours, with 0 (indicating "No pain") and 10 (indicating "Worst pain imaginable). Higher scores indicated worse pain.
Time Frame: At Week 16
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 173 | 88
Percentage of participants | 51.6 | 27.5

10. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Body Surface Area (BSA) at Weeks 2, 4, 8, 12 and 16
Description: The BSA assessment estimates the extent of disease or skin involvement with respect to AD and is expressed as a percentage of total body surface. BSA was determined by the Investigator or designee using the participant palm = 1% BSA rule. The participant's palm is measured from the wrist to the proximal interphalangeal and thumb. This higher the BSA %, the more active atopic dermatitis is present. Percent of BSA for a body region = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA for an individual is arithmetic mean of % BSA of all 4 body regions and ranges from 0% to 100% with higher values representing greater severity of AD and negative change from baseline indicate no severity.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage of body surface area
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 217 | 111
Percentage of body surface area
  Change at Week 2: number analyzed (Participants) | 216 | 111
  Change at Week 2 | -11.4 (15.33) | -10.6 (12.04)
  Change at Week 4: number analyzed (Participants) | 217 | 107
  Change at Week 4 | -19.5 (19.22) | -15.3 (13.77)
  Change at Week 8: number analyzed (Participants) | 211 | 102
  Change at Week 8 | -27.3 (20.60) | -19.2 (17.12)
  Change at Week 12: number analyzed (Participants) | 205 | 99
  Change at Week 12 | -30.6 (21.25) | -22.5 (17.06)
  Change at Week 16: number analyzed (Participants) | 209 | 99
  Change at Week 16 | -32.5 (21.44) | -22.1 (18.57)

11. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) at Weeks 8 and 16
Description: SCORAD is a validated clinical tool for assessing the extent and intensity of AD. There are 3 components: A) Surface involvement is assessed as proportion of involved surface area segment by segment by applying the rule of 9s and reported as the sum of all areas, with a score ranging from 0-100. B) Intensity part of the SCORAD consists of 6 items: erythema, oedema, oozing/crusting, excoriation, lichenification, and dryness. Each item graded as: none (0), mild (1), moderate (2), or severe (3). C) Subjective assessment of itch and of sleeplessness is recorded for each symptom using a visual analogue scale (VAS), where 0=no itch (or no sleeplessness) and 10= worst imaginable itch (or sleeplessness), with maximum score of 20. Formula is: A/5+7B/2+C, A: extent (0-100), B: intensity (0-18), C: subjective symptoms (0-20). SCORAD total score ranged from 0 (no disease) to 103 (severe disease). Higher values represent worse outcome and negative change from baseline indicate improvement.
Time Frame: Baseline, Weeks 8 and 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 199 | 94
Score on a Scale
  Change at Week 8: number analyzed (Participants) | 198 | 94
  Change at Week 8 | -32.1 (17.90) | -20.0 (18.04)
  Change at Week 16: number analyzed (Participants) | 199 | 89
  Change at Week 16 | -36.8 (20.40) | -23.7 (21.25)

12. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Pruritus NRS by Week up to Week 16
Description: The Pruritus NRS is an 11-point scale used by participants to rate their worst pruritus (itch) severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable." Higher scores indicated greater severity and negative change from baseline indicate no severity.
Time Frame: Baseline, Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 214 | 108
Score on a Scale
  Change at Week 2: number analyzed (Participants) | 206 | 105
  Change at Week 2 | -1.543 (1.6304) | -1.113 (1.7468)
  Change at Week 3: number analyzed (Participants) | 213 | 108
  Change at Week 3 | -2.199 (2.0960) | -1.420 (2.1401)
  Change at Week 4: number analyzed (Participants) | 214 | 107
  Change at Week 4 | -2.351 (2.2558) | -1.450 (2.3924)
  Change at Week 5: number analyzed (Participants) | 211 | 101
  Change at Week 5 | -2.771 (2.4152) | -1.485 (2.4553)
  Change at Week 6: number analyzed (Participants) | 207 | 101
  Change at Week 6 | -3.053 (2.3975) | -1.711 (2.5330)
  Change at Week 7: number analyzed (Participants) | 203 | 101
  Change at Week 7 | -3.204 (2.4643) | -1.823 (2.5263)
  Change at Week 8: number analyzed (Participants) | 212 | 99
  Change at Week 8 | -3.080 (2.4552) | -1.856 (2.5670)
  Change at Week 9: number analyzed (Participants) | 205 | 100
  Change at Week 9 | -3.283 (2.5105) | -1.861 (2.5872)
  Change at Week 10: number analyzed (Participants) | 205 | 98
  Change at Week 10 | -3.245 (2.6101) | -1.529 (2.7489)
  Change at Week 11: number analyzed (Participants) | 201 | 96
  Change at Week 11 | -3.285 (2.5484) | -1.776 (2.7302)
  Change at Week 12: number analyzed (Participants) | 206 | 97
  Change at Week 12 | -3.388 (2.6195) | -1.853 (2.3583)
  Change at Week 13: number analyzed (Participants) | 196 | 97
  Change at Week 13 | -3.326 (2.6697) | -2.053 (2.5284)
  Change at Week 14: number analyzed (Participants) | 203 | 96
  Change at Week 14 | -3.313 (2.6843) | -1.948 (2.4181)
  Change at Week 15: number analyzed (Participants) | 202 | 96
  Change at Week 15 | -3.366 (2.5291) | -1.938 (2.5245)
  Change at Week 16: number analyzed (Participants) | 203 | 92
  Change at Week 16 | -3.476 (2.5453) | -2.183 (2.4246)

13. Secondary Outcome: Double-blind Induction Period: Change From Baseline in the Sleep Loss at Week 16 Using Patient-related Outcome (PRO) by Week up to Week 16
Description: Sleep loss was assessed by all participants using a PRO instrument. Participants (and if applicable, with help of parents/caregiver if required) rate their sleep on a 5-point Likert scale (with scores ranging from 0 [not at all] to 4 [unable to sleep at all]). Higher scores indicated a greater impact and worse outcome; therefore, negative change from baseline indicate less impact.
Time Frame: Baseline, Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 214 | 108
Score on a Scale
  Change at Week 2: number analyzed (Participants) | 206 | 105
  Change at Week 2 | -0.603 (0.6985) | -0.493 (0.8407)
  Change at Week 3: number analyzed (Participants) | 213 | 108
  Change at Week 3 | -0.816 (0.8809) | -0.673 (1.0262)
  Change at Week 4: number analyzed (Participants) | 214 | 107
  Change at Week 4 | -0.875 (0.9387) | -0.577 (1.0885)
  Change at Week 5: number analyzed (Participants) | 210 | 101
  Change at Week 5 | -0.942 (0.9646) | -0.607 (1.1342)
  Change at Week 6: number analyzed (Participants) | 207 | 101
  Change at Week 6 | -0.998 (0.9088) | -0.613 (1.0641)
  Change at Week 7: number analyzed (Participants) | 203 | 101
  Change at Week 7 | -1.038 (0.9388) | -0.661 (1.1119)
  Change at Week 8: number analyzed (Participants) | 212 | 99
  Change at Week 8 | -0.974 (0.9941) | -0.708 (1.1500)
  Change at Week 9: number analyzed (Participants) | 205 | 100
  Change at Week 9 | -1.052 (0.9352) | -0.668 (1.0604)
  Change at Week 10: number analyzed (Participants) | 205 | 98
  Change at Week 10 | -1.091 (0.9624) | -0.560 (1.1349)
  Change at Week 11: number analyzed (Participants) | 201 | 96
  Change at Week 11 | -1.040 (0.9966) | -0.676 (1.0938)
  Change at Week 12: number analyzed (Participants) | 206 | 97
  Change at Week 12 | -1.123 (1.0281) | -0.721 (1.0768)
  Change at Week 13: number analyzed (Participants) | 196 | 97
  Change at Week 13 | -1.069 (0.9776) | -0.797 (1.1037)
  Change at Week 14: number analyzed (Participants) | 203 | 96
  Change at Week 14 | -1.072 (1.0446) | -0.809 (1.0751)
  Change at Week 15: number analyzed (Participants) | 202 | 96
  Change at Week 15 | -1.096 (0.9819) | -0.756 (1.0891)
  Change at Week 16: number analyzed (Participants) | 203 | 92
  Change at Week 16 | -1.201 (0.9775) | -0.857 (1.0615)

14. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Patient-Oriented Eczema Measure (POEM) Total Score at Weeks 4, 8, 12 and 16
Description: The POEM is a 7-item, validated questionnaire completed by the participant (and, if applicable, with help of parents/caregiver if required) to assess disease symptoms. Participants are asked to respond to questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping. All answers carry equal weight, with a total possible score ranging from 0 to 28 (answers scored as: No days = 0; 1 to 2 days = 1; 3 to 4 days = 2; 5 to 6 days = 3; every day = 4. Higher scores indicated more severe disease and poor quality of life (QoL); therefore, negative change from baseline indicate improvement in QoL.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 201 | 98
Score on a Scale
  Change at Week 4 | -8.4 (6.82) | -4.7 (6.42)
  Change at Week 8: number analyzed (Participants) | 199 | 91
  Change at Week 8 | -10.9 (7.45) | -5.2 (6.65)
  Change at Week 12: number analyzed (Participants) | 197 | 87
  Change at Week 12 | -11.3 (8.08) | -5.1 (7.25)
  Change at Week 16: number analyzed (Participants) | 196 | 87
  Change at Week 16 | -11.9 (8.01) | -5.8 (7.18)

15. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Weeks 2. 4, 8, 12 and 16
Description: The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question was scored on a 4-point scale (ranged from 0 to 3) where, 0 = not at all, 1= a little, 2= a lot, 3= very much, giving a total score ranging from 0 (not at all) to 30 (very much). A high score is indicative of a poor QoL and negative change from baseline indicate improvement in QoL.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 185 | 91
Score on a Scale
  Change at Week 2 | -4.6 (5.54) | -4.5 (6.00)
  Change at Week 4: number analyzed (Participants) | 178 | 90
  Change at Week 4 | -7.1 (6.54) | -5.4 (6.86)
  Change at Week 8: number analyzed (Participants) | 177 | 83
  Change at Week 8 | -8.3 (7.03) | -5.7 (7.89)
  Change at Week 12: number analyzed (Participants) | 176 | 79
  Change at Week 12 | -8.7 (7.38) | -5.9 (7.90)
  Change at Week 16: number analyzed (Participants) | 175 | 79
  Change at Week 16 | -9.5 (7.40) | -8.1 (7.62)

16. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 2. 4, 8, 12 and 16
Description: The CDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI to measure the impact of AD disease on QoL in children during the previous week. Each question is scored as follows: 0=not at all or unanswered, 1 = only a little, 2 = quite a lot and 3 = very much. Question 7 has an added possible response, which was scored as 3. CDLQI equals the sum of the score of each question, ranged from 0 (no impact of skin disease on QoL) to 30 (maximum impact on QoL). Higher scores indicate higher impact on QoL and negative change from baseline indicate low impact on QoL.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 23 | 8
Score on a Scale
  Change at Week 2 | -2.9 (3.41) | -3.6 (3.25)
  Change at Week 4 | -5.1 (4.76) | -4.3 (4.65)
  Change at Week 8 | -6.6 (6.69) | -6.9 (4.82)
  Change at Week 12: number analyzed (Participants) | 21 | 8
  Change at Week 12 | -7.7 (7.60) | -7.4 (6.30)
  Change at Week 16: number analyzed (Participants) | 21 | 8
  Change at Week 16 | -7.7 (6.91) | -6.8 (5.73)

17. Secondary Outcome: Double-blind Induction Period: Change From Baseline in Skin Pain NRS by Week up to Week 16
Description: The Skin Pain NRS is an 11-point scale completed by participants to rate their worst skin pain (example, discomfort or soreness) severity over the past 24 hours, with 0 (indicating "No pain") to 10 (indicating "Worst pain imaginable). Higher scores indicated worse pain and negative change from baseline indicate no pain.
Time Frame: Baseline, Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 214 | 108
Score on a Scale
  Change at Week 2: number analyzed (Participants) | 206 | 105
  Change at Week 2 | -1.546 (1.7978) | -0.905 (1.9170)
  Change at Week 3: number analyzed (Participants) | 213 | 108
  Change at Week 3 | -2.152 (2.1719) | -1.316 (2.2680)
  Change at Week 4: number analyzed (Participants) | 214 | 107
  Change at Week 4 | -2.308 (2.2457) | -1.271 (2.4880)
  Change at Week 5: number analyzed (Participants) | 211 | 101
  Change at Week 5 | -2.589 (2.3577) | -1.333 (2.4462)
  Change at Week 6: number analyzed (Participants) | 207 | 101
  Change at Week 6 | -2.862 (2.4428) | -1.309 (2.5079)
  Change at Week 7: number analyzed (Participants) | 203 | 101
  Change at Week 7 | -2.886 (2.4473) | -1.656 (2.4816)
  Change at Week 8: number analyzed (Participants) | 212 | 99
  Change at Week 8 | -2.872 (2.4975) | -1.711 (2.7208)
  Change at Week 9: number analyzed (Participants) | 205 | 100
  Change at Week 9 | -3.017 (2.4897) | -1.598 (2.5693)
  Change at Week 10: number analyzed (Participants) | 205 | 98
  Change at Week 10 | -3.017 (2.6017) | -1.382 (2.7463)
  Change at Week 11: number analyzed (Participants) | 201 | 96
  Change at Week 11 | -3.116 (2.6230) | -1.572 (2.6465)
  Change at Week 12: number analyzed (Participants) | 206 | 97
  Change at Week 12 | -3.115 (2.6181) | -1.520 (2.5976)
  Change at Week 13: number analyzed (Participants) | 196 | 97
  Change at Week 13 | -3.140 (2.5568) | -1.788 (2.4726)
  Change at Week 14: number analyzed (Participants) | 203 | 96
  Change at Week 14 | -3.035 (2.6733) | -1.683 (2.4462)
  Change at Week 15: number analyzed (Participants) | 203 | 96
  Change at Week 15 | -3.138 (2.6062) | -1.781 (2.6443)
  Change at Week 16: number analyzed (Participants) | 203 | 92
  Change at Week 16 | -3.302 (2.5844) | -1.831 (2.5766)

18. Secondary Outcome: Double-blind Induction Period: Proportion of Topical Corticosteroids (TCS) Medication Free Days
Description: TCS free days proportion = Number of days participant did not take TCS medication / Number of days from Baseline to Week 16 Date or early discontinuation
Time Frame: Baseline up to Week 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Mean (Standard Deviation); unit: Proportion of Days
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Proportion of Days | 0.224 (0.3491) | 0.151 (0.3032)

19. Secondary Outcome: Double-blind Induction Period: Median Time (Days) to TCS-Free Use
Description: Days from first study drug injection to the day participant stopped using all TCS.
Time Frame: Baseline up to Week 16
Population: FAS included all randomized participants and were analyzed under the treatment group as randomized.
Measure: Median (Full Range); unit: Days
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS
Number analyzed (Participants) | 220 | 111
Days | NA [NA to NA] — Median and full range was not estimated due to insufficient number of events. | NA [NA to NA] — Median and full range was not estimated due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: Double-blind Induction Period: Day 1 to Week 16; Open-label Maintenance Period: Week 16 to Week 52
Arm/Group | Double-blind Induction Period: Lebrikizumab +TCS | Double-blind Induction Period: Placebo +TCS | Open-label Maintenance Period: Lebrikizumab to Lebrikizumab | Open-label Maintenance Period: Placebo to Lebrikizumab
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/111 | 0/212 | 0/100
Serious Adverse Events (participants affected / at risk) | 3/220 | 1/111 | 12/212 | 4/100
Other Adverse Events (participants affected / at risk) | 84/220 | 31/111 | 108/212 | 48/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Induction Period: Lebrikizumab +TCS (N=220) | Double-blind Induction Period: Placebo +TCS (N=111) | Open-label Maintenance Period: Lebrikizumab to Lebrikizumab (N=212) | Open-label Maintenance Period: Placebo to Lebrikizumab (N=100)
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Induction Period: Lebrikizumab +TCS (N=220) | Double-blind Induction Period: Placebo +TCS (N=111) | Open-label Maintenance Period: Lebrikizumab to Lebrikizumab (N=212) | Open-label Maintenance Period: Placebo to Lebrikizumab (N=100)
Conjunctivitis allergic (Eye disorders) | 18 | 3 | 18 | 11
COVID-19 (Infections and infestations) | 8 | 7 | 13 | 4
Conjunctivitis (Infections and infestations) | 25 | 2 | 25 | 11
Nasopharyngitis (Infections and infestations) | 28 | 14 | 52 | 16
Oral herpes (Infections and infestations) | 11 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 17 | 6
Headache (Nervous system disorders) | 6 | 6 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05149313/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05149313/SAP_001.pdf